CLINICAL TRIAL: NCT04702113
Title: Evaluating Pharmacogenomic Variants for Cardiology Therapeutics: the Lighthouse Pilot (Association Between Genetic Variant Scores and P2Y12 Inhibitor Effects)
Brief Title: Evaluating Pharmacogenomic Variants for Cardiology Therapeutics
Acronym: CARES2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cipherome, Inc. (Industry)
Collaborators: DHR Health Institute for Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: C03-002 DHR001
Record Dates: First submitted 2020-12-14; First posted 2021-01-08 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Thrombosis; Stent Thrombosis; Bleeding; Myocardial Infarction; Ischemic Stroke
Keywords: Stent Thrombosis; Major Adverse Cardiovascular and Cerebrovascular Events (MACCE)
MeSH Terms: conditions — Thrombosis; Hemorrhage; Myocardial Infarction; Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: There will be two study arms:
  1. Conventional therapy (controls)-treatment with clopidogrel and no pre-emptive genotyping
  2. Genotype-guided therapy (experimental)
Masking Description: This is an open label study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Therapy (Controls) (No Intervention): Treatment with clopidogrel and no pre-emptive genotyping
- Genotype-guided therapy (experimental) (Experimental): 1. Treatment with clopidogrel 75 mg daily for non-carriers
  2. Treatment with ticagrelor 90 mg twice daily for carriers
  Interventions: Diagnostic Test: Cipherome Lighthouse Pilot

INTERVENTIONS:
Diagnostic Test: Cipherome Lighthouse Pilot — Preemptive pharmacogenomic testing
  Arms: Genotype-guided therapy (experimental)

SUMMARY:
Cipherome's Lighthouse is a clinical decision support tool that incorporates a patient's pharmacogenetic information to determine therapeutic strategy, including determining appropriate dosage or assessing the likelihood of toxicity of a therapeutic regimen.

DETAILED DESCRIPTION:
The Lighthouse tool incorporates pharmacogenetic (PGx) variants from well-established, evidence-based guidelines to provide personalized drug response profile(s) to guide treatment decisions.

The patient specimen is genotyped using a proprietary, carefully curated pharmacogenetic variant panel to determine the individual's phenotype. The Lighthouse report (PGx findings) are provided to the clinician, and a notification is generated when the patient has a genotype with a deleterious drug-metabolizing phenotype.

Evaluating the South Texas community for the pilot project will enhance the understanding of the impact of genetic variants on individuals of Hispanic/Latino ancestry, especially as the variants pertain to the efficacy and safety of medications.

ELIGIBILITY:
Inclusion Criteria:

* Subjects over 18 years of age, who are:
* On clopidogrel, prasugrel or ticagrelor after percutaneous stent
* Completed informed consent

Exclusion Criteria:

* Failure to provide informed consent.
* Lost to follow-up prior to 60 days.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2020-12-03 (Actual); Primary Completion 2023-07-26 (Actual); Study Completion 2023-07-27 (Actual)

PRIMARY OUTCOMES:
Evaluation of aggregate costs | Study pilot duration is 365 days (1 year)
  The cumulative direct medical cost (admissions, procedures, clinical visits, blood transfusions, drugs) of percutaneous insertion of stents (PCIs) and associated major adverse cardiovascular and cerebrovascular events (MACCE) including non-fatal myocardial infarction, non-fatal stroke, cardiovascular mortality, severe recurrent ischemia and stent thrombosis, and the costs of P2Y12 inhibitors and pharmacogenomic test costs.

SECONDARY OUTCOMES:
Reduction of treatment failures | Study pilot duration is 365 days (1 year)
  Reduced treatment failures within 30, 60, 90 days, and 12 months of receiving clopidogrel in participants with reduced function alleles (CYP2C19 *2 or *3)
Reduction of major or minor bleeding events | Study pilot duration is 365 days (1 year)
  Reduced major or minor bleeding events within 30, 60, 90 days, and 12 months of receiving clopidogrel in participants with increased function alleles (CYP2C19 *17)

OTHER OUTCOMES:
Assessment of the correlation of clinical factors (age, labs, medications) on predicting and preventing adverse drug reactions | Study pilot duration is 365 days (1 year)
  Assess the correlation of clinical factors (age, liver function tests, concomitant medications, etc.) on predicting and preventing adverse drug reactions (ADRs).

CONTACTS AND LOCATIONS:
Overall Officials: Herschl Silberman, MD, Principal Investigator — DHR Health; Humberto Mochizu Kitamayo, MD, Study Director — DHR Health; Yetunde O Kare Opaneye, MD, Study Director — DHR Health
Locations (1):
- Doctors Hospital at Renaissance, Edinburg, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Claudio-Campos K, Duconge J, Cadilla CL, Ruano G. Pharmacogenetics of drug-metabolizing enzymes in US Hispanics. Drug Metab Pers Ther. 2015 Jun;30(2):87-105. doi: 10.1515/dmdi-2014-0023. PMID 25431893
- [Background] Dean L, Kane M. Prasugrel Therapy and CYP Genotype. 2017 Apr 10 [updated 2024 Oct 15]. In: Pratt VM, Scott SA, Pirmohamed M, Esquivel B, Kattman BL, Malheiro AJ, editors. Medical Genetics Summaries [Internet]. Bethesda (MD): National Center for Biotechnology Information (US); 2012-. Available from http://www.ncbi.nlm.nih.gov/books/NBK425796/ PMID 28520385
- [Background] Lee CR, Sriramoju VB, Cervantes A, Howell LA, Varunok N, Madan S, Hamrick K, Polasek MJ, Lee JA, Clarke M, Cicci JD, Weck KE, Stouffer GA. Clinical Outcomes and Sustainability of Using CYP2C19 Genotype-Guided Antiplatelet Therapy After Percutaneous Coronary Intervention. Circ Genom Precis Med. 2018 Apr;11(4):e002069. doi: 10.1161/CIRCGEN.117.002069. PMID 29615454
- [Background] Levine GN, Bates ER, Bittl JA, Brindis RG, Fihn SD, Fleisher LA, Granger CB, Lange RA, Mack MJ, Mauri L, Mehran R, Mukherjee D, Newby LK, O'Gara PT, Sabatine MS, Smith PK, Smith SC Jr, Halperin JL, Levine GN, Al-Khatib SM, Birtcher KK, Bozkurt B, Brindis RG, Cigarroa JE, Curtis LH, Fleisher LA, Gentile F, Gidding S, Hlatky MA, Ikonomidis JS, Joglar JA, Pressler SJ, Wijeysundera DN. 2016 ACC/AHA guideline focused update on duration of dual antiplatelet therapy in patients with coronary artery disease: A report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. J Thorac Cardiovasc Surg. 2016 Nov;152(5):1243-1275. doi: 10.1016/j.jtcvs.2016.07.044. No abstract available. PMID 27751237
- [Background] Limdi NA, Cavallari LH, Lee CR, Hillegass WB, Holmes AM, Skaar TC, Pisu M, Dillon C, Beitelshees AL, Empey PE, Duarte JD, Diaby V, Gong Y, Johnson JA, Graves J, Garbett S, Zhou Z, Peterson JF; Implementing GeNomics In pracTicE (IGNITE) Network Pharmacogenetic Working Group (IGNITE-PGx). Cost-effectiveness of CYP2C19-guided antiplatelet therapy in patients with acute coronary syndrome and percutaneous coronary intervention informed by real-world data. Pharmacogenomics J. 2020 Oct;20(5):724-735. doi: 10.1038/s41397-020-0162-5. Epub 2020 Feb 11. PMID 32042096
- [Background] Mega JL, Simon T, Collet JP, Anderson JL, Antman EM, Bliden K, Cannon CP, Danchin N, Giusti B, Gurbel P, Horne BD, Hulot JS, Kastrati A, Montalescot G, Neumann FJ, Shen L, Sibbing D, Steg PG, Trenk D, Wiviott SD, Sabatine MS. Reduced-function CYP2C19 genotype and risk of adverse clinical outcomes among patients treated with clopidogrel predominantly for PCI: a meta-analysis. JAMA. 2010 Oct 27;304(16):1821-30. doi: 10.1001/jama.2010.1543. PMID 20978260
- [Background] Mehran R, Rao SV, Bhatt DL, Gibson CM, Caixeta A, Eikelboom J, Kaul S, Wiviott SD, Menon V, Nikolsky E, Serebruany V, Valgimigli M, Vranckx P, Taggart D, Sabik JF, Cutlip DE, Krucoff MW, Ohman EM, Steg PG, White H. Standardized bleeding definitions for cardiovascular clinical trials: a consensus report from the Bleeding Academic Research Consortium. Circulation. 2011 Jun 14;123(23):2736-47. doi: 10.1161/CIRCULATIONAHA.110.009449. No abstract available. PMID 21670242
- [Background] Parks AL, Fang MC. Scoring Systems for Estimating the Risk of Anticoagulant-Associated Bleeding. Semin Thromb Hemost. 2017 Jul;43(5):514-524. doi: 10.1055/s-0037-1598061. Epub 2017 Mar 30. PMID 28359135
- [Background] Pereira NL, Farkouh ME, So D, Lennon R, Geller N, Mathew V, Bell M, Bae JH, Jeong MH, Chavez I, Gordon P, Abbott JD, Cagin C, Baudhuin L, Fu YP, Goodman SG, Hasan A, Iturriaga E, Lerman A, Sidhu M, Tanguay JF, Wang L, Weinshilboum R, Welsh R, Rosenberg Y, Bailey K, Rihal C. Effect of Genotype-Guided Oral P2Y12 Inhibitor Selection vs Conventional Clopidogrel Therapy on Ischemic Outcomes After Percutaneous Coronary Intervention: The TAILOR-PCI Randomized Clinical Trial. JAMA. 2020 Aug 25;324(8):761-771. doi: 10.1001/jama.2020.12443. PMID 32840598
- [Background] Wasfy JH, Strom JB, Waldo SW, O'Brien C, Wimmer NJ, Zai AH, Luttrell J, Spertus JA, Kennedy KF, Normand SL, Mauri L, Yeh RW. Clinical preventability of 30-day readmission after percutaneous coronary intervention. J Am Heart Assoc. 2014 Sep 26;3(5):e001290. doi: 10.1161/JAHA.114.001290. PMID 25261531
- [Background] MEPS 2019. Agency for Healthcare Research and Quality. Medical Expenditure Panel Survey. MEPS HC-197A: 2017. Prescribed Medicines File. July 2019.
- [Background] Pereira NL, Rihal CS, So DYF, Rosenberg Y, Lennon RJ, Mathew V, Goodman SG, Weinshilboum RM, Wang L, Baudhuin LM, Lerman A, Hasan A, Iturriaga E, Fu YP, Geller N, Bailey K, Farkouh ME. Clopidogrel Pharmacogenetics. Circ Cardiovasc Interv. 2019 Apr;12(4):e007811. doi: 10.1161/CIRCINTERVENTIONS.119.007811. PMID 30998396
- [Background] Pereira INTV 2020. CC News Story, TAILOR-PCI: Genotype-guided Antiplatelet Therapy Post PCI Misses Mark. American Academy of Cardiology. Pulled 18 September 2020. https://www.acc.org/latest-in-cardiology/articles/2020/03/24/16/41/sat-9am-tailor-pci-clinical-implementation-clopidogrel-pharmacogenetics-acc-2020.
- [Background] Python 2020. Python code Mersenne Twister core generator with a period of (219937 -1). The Python Standard Library / Numeric and Mathematical Modules / random - Generate pseudo-random numbers. https://docs.python.org/3/library/random.html
- [Background] Yost GW, Puher SL, Graham J, Scott TD, Skelding KA, Berger PB, Blankenship JC. Readmission in the 30 days after percutaneous coronary intervention. JACC Cardiovasc Interv. 2013 Mar;6(3):237-44. doi: 10.1016/j.jcin.2012.10.015. PMID 23517834
- See also: Clinical Pharmacogenetics Implementation Consortium (CPIC) 2020 — https://www.fda.gov/medical-devices/precision-medicine/table-pharmacogenetic-associations
- See also: FDA ADR 2020 — https://fis.fda.gov/sense/app/d10be6bb-494e-4cd2-82e4-0135608ddc13/sheet/7a47a261-d58b-4203-a8aa-6d3021737452/state/analysis
- See also: FDA ADR 2020 — https://data.worldbank.org/indicator/SP.POP.TOTL?locations=US
- See also: Sauer 2017. PCI Within the Context of the Episode Payment Model — https://citoday.com/articles/2017-sept-oct/pci-within-the-context-of-the-episode-payment-model
- See also: Simmons 2018. Clearwater Corporation, "Letter to HHS Physician Focused Payment Model Technical Advisory Committee" — https://aspe.hhs.gov/system/files/pdf/255906/ProposalClearwater.pdf
- See also: Truesdale 2017. Truesdale K., Corazon, Inc. "Change is coming in 2018-be prepared! — https://citoday.com/articles/2017-sept-oct/pci-within-the-context-of-the-episode-payment-model
- See also: Change is coming in 2018-be prepared! — https://citoday.com/articles/2017-sept-oct/pci-within-the-context-of-the-episode-payment-model
- See also: TAILOR PCI — https://clinicaltrials.gov/ct2/show/NCT01742117?term=TAILOR+PCI&rank=1
- See also: TAILOR PCI — https://www.acc.org/latest-in-cardiology/articles/2020/03/24/16/41/sat-9am-tailor-pci-clinical-implementation-clopidogrel-pharmacogenetics-acc-2020